CLINICAL TRIAL: NCT06601075
Title: The Role of 18F-FDG and 68Ga-FAPI PET/CT in the Diagnosis and the Efficacy Evaluation of Advanced Colorectal Cancer (peritoneal Metastasis With/without Other Metastases)
Status: Recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Hu Jiajia, Deputy director, Ruijin Hospital
Other Study IDs: RuijinH 2024-80
Record Dates: First submitted 2024-09-14; First posted 2024-09-19 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Advanced Colorectal Cancer
Keywords: 68Ga-FAPI PET/CT; diagnosis; advanced colorectal cancer; efficacy evaluation
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients diagnosis of advanced colorectal cancer: Patients diagnosis of advanced colorectal cancer (peritoneal metastasis with/without other metastases)

SUMMARY:
This study aims to investigate the value of 18F-FDG and 68Ga-FAPI PET/CT in evaluating the outcome of conversion therapy and the prognosis of advanced colorectal cancer (peritoneal metastasis with/without other metastases)

DETAILED DESCRIPTION:
The investigators will number all participants, create a medical record file, and record their basic information (gender, age) as well as contact information and medical history information. All participants will undergo 18F-FDG and 68Ga-FAPI PET/CT at baseline and after 3 months of conversion therapy. The imaging response measurements will be compared with the histopathological or clinical assessment results as gold standard.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed colorectal cancer, clinical or other imaging suspicion of peritoneal metastasis with or without other distant metastases.
2. Patients voluntarily enrolled in this study by signing an informed consent form
3. Age ≥ 18 years
4. Expected life expectancy ≥ 3 months
5. Adequate organ and bone marrow function
6. Willingness to adhere to the study protocol and follow-up programme

Exclusion Criteria:

1. Pregnant or breastfeeding women.
2. Patients with a history of other malignant diseases in the last 5 years, except cured skin cancer and carcinoma in situ of cervix
3. Severe mental disease, uncontrolled epilepsy, or central nervous system disease
4. Subjects with current concurrent interstitial pneumonitis or interstitial lung disease, or subjects with previous interstitial pneumonitis or interstitial lung disease requiring hormonal therapy, or subjects with other conditions that may interfere with the judgement and management of immune-related pulmonary toxicity, e.g., pulmonary fibrosis, organising pneumonia (e.g., occlusive bronchiectasis), pulmonary fibrosis, organising pneumonia (e.g., occlusive bronchiectasis), pneumoconiosis, Drug-associated pneumonia, idiopathic pneumonia, active pneumonia, or severe pulmonary impairment on CT; and active tuberculosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible inpatients and outpatients from Ruijin Hospital
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy | Baseline and up to 3 months
  18F-FDG and 68Ga-FAPI PET/CT was used to diagnose the lesions of the patients, and the diagnostic performance of PET/CT was evaluated by comparing the diagnostic results with the pathological results/clinical evaluation results.
Standardized uptake value(SUV) | Baseline and up to 3 months
  SUV of 68Ga-FAPI and 18F-FDG uptake on PET/CT images for tumor lesions
Target-to-background ratio(TBR) | Baseline and up to 3 months
  68Ga-FAPI and 18F-FDG uptake ratio of tumor lesions to mediastinum and liver blood pool on PET/CT images.

SECONDARY OUTCOMES:
Progress free survival | 3 years
  Progress free survival
Overall survival | 3 years
  Overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital affiliated to Shanghai Jiao Tong University of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No